CLINICAL TRIAL: NCT00572481
Title: ARM: Axillary Reverse Mapping, A Prospective Study
Brief Title: Axillary Reverse Mapping
Acronym: ARM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 78076
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Cancer of the Breast
Keywords: Sentinel Lymph Node Biopsy; Axillary Node Dissection; Prevention of lymphedema; Prevention of neuroma; Prevention of seroma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: During surgery, the technetium-99m sulfur colloid will be injected into the breast and the blue dye injected (if the patient is not allergic and it is not required to locate the SLN) in the patient's ipsilateral upper arm. The lymph node biopsy and/or dissection will be performed by the surgeon, according to standard practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sentinel Lymph Node Biopsy Only (Other): Axillary Reverse Mapping
  Interventions: Procedure: Axillary Reverse Mapping
- Full Axillary Lymph Node Dissection (Other): Axillary Reverse Mapping
  Interventions: Procedure: Axillary Reverse Mapping

INTERVENTIONS:
Procedure: Axillary Reverse Mapping — During surgery, the technetium-99m sulfur colloid will be injected into the breast and the blue dye injected (if the patient is not allergic and it is not required to locate the SLN) in the patient's ipsilateral upper arm. The lymph node biopsy and/or dissection will be performed by the surgeon, according to standard practice.

SUMMARY:
We hypothesize that variations in anatomic location of the arm lymphatic drainage system put the arm lymphatics at risk for disruption during a SLNB and / or ALND. Therefore, mapping the drainage of the arm during the procedure would decrease the likelihood of inadvertent disruption of the lymphatics and the subsequent development of lymphedema. A combination of radioactivity and blue dye will be used.

DETAILED DESCRIPTION:
Mapping Procedure:

Each patient will receive an injection of 1.0 mCi of technetium-99m sulfur colloid into the normal breast tissue surrounding the primary cancer or biopsy cavity directed subareolar or around the tumor.

If the radioactive SLN cannot be located prior to incision via gamma probe then the blue dye will be used in the breast either in the subareolar plexus or peritumorally at the discretion of the surgeon. For this contingency (expected to occur <3% of the time), the blue dye will be used in the breast (and NOT the arm), as the prime concern is locating the SLN for staging.

If the blue dye is unnecessary to find the sentinel node draining from the breast, then it will be injected dermally in the upper inner arm along the Biceps groove of the ipsilateral arm in order to locate the draining lymphatics from the arm. No more than 5cc of blue dye will be injected in either the subareolar plexus, peritumorally (intraparenchymal or dermally), or dermally in the patient's ipsilateral arm dependent upon the contingencies stated above. Site of all injections (radioactivity and/or blue dye) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-100 years old
* Not pregnant or breastfeeding
* Breast cancer requiring lymph node evaluation for the ipsilateral or contralateral breast OR prophylactic mastectomy
* Willing participation following an informed consent process

Exclusion Criteria:

* Patient < 18 y/o or > 100 y/o
* Pregnant or breastfeeding
* If a pregnant female should be diagnosed with breast cancer an exception would be considered on a case to case basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Occurrence of lymphedema by the first year following surgery | One year
  An occurrence will consist of an increase of 20% or more in ipsilateral arm volume over the pre-surgery volume, and be accompanied by a confirmatory diagnosis of lymphedema from the UAMS lymphedema clinic.

SECONDARY OUTCOMES:
Successful identification (i.e., localization) of breast SLN and arm lymphatics | Time of surgery
  successful localization of one or more lymph nodes to which the peritumoral breast region drains
Characterization of location (typical versus variant) of arm lymphatics. | Time of surgery
  brief location details will also be collected.
Successful protection of the arm lymphatics during SLNB and/or ALND. | Time of surgery
  successful avoidance of resection and/or successful preservation of structural integrity of arm lymphatics during the surgical procedure.
Occurrence of crossover (i.e., co-localization) between hot breast SLN and blue arm lymphatics. | Time of surgery
  A crossover event will consist of identification of one or more lymph nodes that are both focally radioactive following peritumoral Tc99m injection and noticeably stained blue following ipsilateral arm injection with Lymphazurin.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ochoa, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas For Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson M, Korourian S, Henry-Tillman R, Adkins L, Mumford S, Westbrook KC, Klimberg VS. Axillary reverse mapping (ARM): a new concept to identify and enhance lymphatic preservation. Ann Surg Oncol. 2007 Jun;14(6):1890-5. doi: 10.1245/s10434-007-9412-x. Epub 2007 May 4. PMID 17479341
- [Background] Klimberg VS. A new concept toward the prevention of lymphedema: axillary reverse mapping. J Surg Oncol. 2008 Jun 1;97(7):563-4. doi: 10.1002/jso.20905. No abstract available. PMID 17955452
- [Result] Boneti C, Korourian S, Bland K, Cox K, Adkins LL, Henry-Tillman RS, Klimberg VS. Axillary reverse mapping: mapping and preserving arm lymphatics may be important in preventing lymphedema during sentinel lymph node biopsy. J Am Coll Surg. 2008 May;206(5):1038-42; discussion 1042-4. doi: 10.1016/j.jamcollsurg.2007.12.022. Epub 2008 Mar 3. PMID 18471751
- [Result] Boneti C, Korourian S, Diaz Z, Santiago C, Mumford S, Adkins L, Klimberg VS. Scientific Impact Award: Axillary reverse mapping (ARM) to identify and protect lymphatics draining the arm during axillary lymphadenectomy. Am J Surg. 2009 Oct;198(4):482-7. doi: 10.1016/j.amjsurg.2009.06.008. PMID 19800452
- [Result] Boneti C, Badgwell B, Robertson Y, Korourian S, Adkins L, Klimberg V. Axillary reverse mapping (ARM): initial results of phase II trial in preventing lymphedema after lymphadenectomy. Minerva Ginecol. 2012 Oct;64(5):421-30. PMID 23018481